CLINICAL TRIAL: NCT02072291
Title: The Influence of Nifedipine Treatment on Uterine Contractility During Frozen Embryo Transfer
Brief Title: Nifedipine Treatment on Uterine Contractility in IVF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nifedipine-FET
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Embryo Implantation
MeSH Terms: interventions — Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nifedipine (Experimental): Nifedipine 5mg single dose
  Interventions: Drug: Nifedipine
- Placebo (Placebo Comparator)
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Nifedipine — PO Nifedipine 5mg single dose

SUMMARY:
The main factors associated with pregnancy rate in In Vitro Fertilization (IVF) treatment are embryo quality and the uterine ability to accept the embryo for implantation. This ability is influenced by uterine contractions (UC), which change in pattern and direction during the menstrual cycle. An abnormal uterine contraction pattern can displace the embryo from the proper position in the uterine cavity towards the cervix or the fallopian tubes and as a result may decrease pregnancy rates and increase the risk of ectopic pregnancy. Indeed, previous studies demonstrated a negative correlation between uterine contraction rate and implantation/pregnancy rates. Suppression of uterine contractions during embryo transfer can be achieved by a large array of drugs, such as cyclo-oxygenase inhibitors, β2-adrenoreceptor agonists, calcium-channel blockers, phosphodiesterase inhibitors and oxytocin antagonists. The objective of this study is to evaluate the efficacy of Nifedipine administration in reducing uterine contractility during IVF-frozen embryo transfer (FET) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing frozen embryo transfer

Exclusion Criteria:

* Body mass index (BMI) > 38 kg/m2
* Early follicular phase (day 2-4) serum follicle stimulating hormone (FSH) level > 20 mIU/ml.
* Abnormal uterine cavity as evidenced by sonohysterogram or hysterosalpingography
* Any contraindication to being pregnant and carrying a pregnancy to term.
* Contraindication for the use of nifedipine, Estrogen and Progesterone suppositories.
* Patient treating with other drugs that interact with cytochrome P450 activity: azole antifungals, cimetidine, cyclosporine, erythromycin, quinidine, terfenadine, warfarin, benzodiazepines, flecainide, imipramine, propafenone and theophylline.
* Irregular heart beat or already being treated with another medication for high blood pressure.
* Any ovarian or abdominal abnormality that may interfere with adequate transvaginal sonography (TVS) evaluation.
* Administration of any investigational drugs within three months prior to study enrollment.
* Patient not able to communicate adequately with the investigators and to comply with the requirements of the entire study.
* Unwillingness to give written informed consent. Previous entry into this study or simultaneous participation in another clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
uterine contractility after treatment | 30 minutes after treatment
  Uterine contractility will be measured by vaginal ultrasound before and 30 minutes after treatment with Nifedipine or placebo

SECONDARY OUTCOMES:
Implantation and pregnancy rates | 4 weeks
  Rates of implantation and clinical pregnancy (cardiac activity) after treatment against placebo

CONTACTS AND LOCATIONS:
Overall Officials: Assaf Ben-Meir, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel